CLINICAL TRIAL: NCT07146022
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Dose Study to Evaluate the Efficacy and Safety of VDPHL01 in Female Subjects With Androgenetic Alopecia
Brief Title: Safety and Efficacy of VDPHL01 in Females With Androgenetic Alopecia (AGA)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Veradermics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250-13951-306
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Androgenetic Alopecia (AGA); Androgenetic Alopecia; AGA; Female Androgenetic Alopecia; Hair Loss
Keywords: Androgenetic Alopecia; AGA; Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VDPHL01 BID (Experimental): VDPHL01 will be taken orally twice a day (BID), once in the AM and once in the PM for the first 6 months of the study. After month 6, subject will continue VDPHL01 BID for an additional 6 months.
  Interventions: Drug: VDPHL01 BID
- VDPHL01 QD and Placebo QD (Experimental): Placebo will be taken orally once a day (QD) in the AM or PM. VDPHL01 will be taken orally once a day (QD) in the AM or PM for the first 6 months of the study. After month 6, subject will continue this same dose regimen for an additional 6 months.
  Interventions: Drug: VDPHL01 QD; Drug: Placebo
- Placebo BID with treatment extension to VDPHL01 BID (Placebo Comparator): Placebo will be taken orally twice a day (BID), once in the AM and once in the PM for the first 6 months of the study. After month 6, subject will switch to VDPHL01 BID group, and take VDPHL01 orally twice a day (BID), once in the AM and once in the PM for an additional 6 months.
  Interventions: Drug: Placebo
- Placebo BID with treatment extension to VDPHL01 QD and Placebo QD (Placebo Comparator): Placebo will be taken orally twice a day (BID), once in the AM and once in the PM for the first 6 months of the study. After month 6, subject will switch to VDPHL01 QD and Placebo QD group, and take placebo orally once a day in the AM or PM; VDPHL01 will be taken orally once a day in the AM or PM for an additional 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VDPHL01 QD — VDPHL01 Extended Release (ER) Tablet
  Arms: VDPHL01 QD and Placebo QD
Drug: Placebo — Placebo tablet
  Arms: Placebo BID with treatment extension to VDPHL01 BID; Placebo BID with treatment extension to VDPHL01 QD and Placebo QD; VDPHL01 QD and Placebo QD
Drug: VDPHL01 BID — VDPHL01 Extended Release (ER) Tablet
  Arms: VDPHL01 BID
Drug: Placebo — Placebo tablet
  Arms: Placebo BID with treatment extension to VDPHL01 BID; Placebo BID with treatment extension to VDPHL01 QD and Placebo QD

SUMMARY:
This study will evaluate the safety and efficacy of VDPHL01 in female subjects with Androgenetic Alopecia (AGA).

AGA is a genetic disorder caused by an excessive (too much) hair follicle response to androgens (hormones) that causes hair loss. VDPHL01 is an investigational oral drug to treat AGA.

This multi-center, double blind, study will last about 13 months and includes 11 study visits (screening, baseline (day 1), week 2, month 1, month 2, month 4, month 6, month 8, month 10, month 12, month 13).

DETAILED DESCRIPTION:
Not required.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female aged 18-65 years old;
* Subject has a clinical diagnosis of mild to moderate AGA;
* Subject is in good general health and has adequate renal and hepatic function;
* Subject is willing to maintain at least 1/4 inch length hair during the study with the same hairstyle, hair length, and hair color throughout the study; maintain consistent use of general hair care products and regimen through the entire study;
* Subject is willing and able to administer the test article as directed and can read, understand, and complete the required questionnaires in English;
* Subject is willing and able to swallow study drug whole;
* Subject agrees to have a micro dot tattoo placed on their scalp;
* Subject agrees to have this area photographed at study visits as indicated in the protocol.

Exclusion Criteria:

* Subject has uncontrolled blood pressure or orthostatic hypotension;
* Subject has symptoms or history of certain heart or thyroid conditions;
* Subject has a history of or active hair loss due to conditions/diseases other than AGA;
* Subject has a current or recent history of dietary or weight changes, including use of GLP-1 agonists;
* Subject has been diagnosed with COVID-19 within 16 weeks of baseline;
* Subject has had previous radiation of the scalp;
* Use of any of the following treatments within the indicated washout period before screening:

  * Subject has used hormone replacement therapy or hormonal modulators within 6 months prior to screening
  * Subject has used oral treatments for hair growth or that can affect hair growth, including systemic retinoids, within 6 months of screening
  * Subject has used systemic calcium channel blockers or beta blockers within 12 weeks prior to screening
  * Subject has used systemic cimetidine, ketoconazole, diazoxide, or corticosteroids (including intramuscular, intraarticular, and intralesional injections) within 12 weeks prior to screening
  * Subject has had any scalp procedures, including surgical, laser, light or energy treatments, micro-needling, injections, platelet rich plasma within 6 months prior to screening
  * Subject has used any topical scalp treatments for hair growth within 12 weeks prior to screening
  * Subject has used any other therapy with any medication either topical or oral that might, in the investigator's opinion, interfere with the study;
  * Subject has any other condition that, in the investigator's opinion, interfere with the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 552 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Changes in non-vellus Target Area Hair Counts (TAHC) | Month 6
  Changes from baseline in non-vellus TAHC using digital image analysis at Month 6.
Subjects Evaluation of Treatment Benefit | Month 6
  Subjects will rate their treatment benefit by responding to a hair assessment scale. The proportion of subjects by each response category will be reported at Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Reid Waldman, M.D., Study Chair — Veradermics, Inc.; Timothy Durso, M.D., Study Chair — Veradermics, Inc.
Locations (71):
- United States (71):
  - Site 73, Birmingham, Alabama
  - Site 89, Birmingham, Alabama
  - Site 77, Phoenix, Arizona
  - Site 30, Fort Smith, Arkansas
  - Site 69, Encino, California
  - Site 2, Fremont, California
  - Site 64, Manhattan Beach, California
  - Site 93, Northridge, California
  - Site 66, Santa Monica, California
  - Site 34, Sherman Oaks, California
  - Site 94, Thousand Oaks, California
  - Site 21, Vista, California
  - Site 5, Castle Rock, Colorado
  - Site 24, Greenwood Village, Colorado
  - Site 17, Aventura, Florida
  - Site 71, Boca Raton, Florida
  - Site 86, Coral Gables, Florida
  - Site 62, Coral Gables, Florida
  - Site 99, Miami, Florida
  - Site 54, Ocala, Florida
  - Site 43, Atlanta, Georgia
  - Site 90, Sandy Springs, Georgia
  - Site 31, Boise, Idaho
  - Site 61, Chicago, Illinois
  - Site 53, Clarksville, Indiana
  - Site 15, Indianapolis, Indiana
  - Site 32, New Albany, Indiana
  - Site 55, Plainfield, Indiana
  - Site 27, West Lafayette, Indiana
  - Site 79, Leawood, Kansas
  - Site 52, Louisville, Kentucky
  - Site 41, Baton Rouge, Louisiana
  - Site 13, Covington, Louisiana
  - Site 12, Metairie, Louisiana
  - Site 75, New Orleans, Louisiana
  - Site 84, Glenn Dale, Maryland
  - Site 87, Rockville, Maryland
  - Site 22, Brighton, Massachusetts
  - Site 80, Chestnut Hill, Massachusetts
  - Site 59, Quincy, Massachusetts
  - Site 26, Clarkston, Michigan
  - Site 68, Clinton Township, Michigan
  - Site 83, Southfield, Michigan
  - Site 98, Medina, Minnesota
  - Site 56, Minneapolis, Minnesota
  - Site 6, New Brighton, Minnesota
  - Site 18, Hackensack, New Jersey
  - Site 37, Kew Gardens, New York
  - Site 97, New York, New York
  - Site 82, Hickory, North Carolina
  - Site 92, Huntersville, North Carolina
  - Site 39, Boardman, Ohio
  - Site 72, Cincinnati, Ohio
  - Site 11, Columbus, Ohio
  - Site 57, Portland, Oregon
  - Site 60, Anderson, South Carolina
  - Site 95, Hermitage, Tennessee
  - Site 9, Knoxville, Tennessee
  - Site 4, Nashville, Tennessee
  - Site 76, Austin, Texas
  - Site 74, College Station, Texas
  - Site 67, Dallas, Texas
  - Site 14, Houston, Texas
  - Site 88, San Antonio, Texas
  - Site 91, Sugar Land, Texas
  - Site 19, South Jordan, Utah
  - Site 29, Forest, Virginia
  - Site 63, Norfolk, Virginia
  - Site 85, Norfolk, Virginia
  - Site 33, Burien, Washington
  - Site 70, Mill Creek, Washington

IPD SHARING:
Plan to Share IPD: Undecided
The sponsor is undecided if this information will be shared at this time. This field will be updated when a decision is made.

REFERENCES:
- See also: Related Info — https://www.phlstudy.com/female/